CLINICAL TRIAL: NCT07257588
Title: Analysis of the Efficacy of Hyperbaric Oxygen-assisted Treatment for Acute Severe Ulcerative Colitis and Refractory Inflammatory Bowel Disease: A Randomized Controlled Study
Brief Title: The Efficacy of Hyperbaric Oxygen-assisted Treatment for ASUC and Refractory IBD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Jie Liang, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJS20242001-C-1
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis
Keywords: Acute severe ulcerative colitis; Refractory inflammatory bowel disease; Heperbaric oxygen-assisted treatment; Randomized controlled study
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heperbaric oxygen-assisted Treatment (Active Comparator): During the 7-day continuous intravenous administration of methylprednisolone sodium succinate at a dose of 40mg per day, hyperbaric oxygen therapy was also provided. The procedure was as follows:
  1. Pressurization: It took 25 minutes to increase the pressure from 1ATA to 2.5ATA (without oxygen inhalation)
  2. Stabilization: A total of 80 minutes (30 minutes of oxygen inhalation, 5 minutes of rest, 30 minutes of oxygen inhalation, 5 minutes of rest, 10 minutes of oxygen inhalation)
  3. Decompression: 25 minutes (the first 18 minutes continued oxygen inhalation, and then 7 minutes of oxygen inhalation was stopped)
  Interventions: Drug: Administration of methylprednisolone sodium succinate; Procedure: Hyperbaric Oxygen Therapy
- Control Treatment (Other): the 7-day continuous intravenous administration of methylprednisolone sodium succinate at a dose of 40mg per day
  Interventions: Drug: Administration of methylprednisolone sodium succinate

INTERVENTIONS:
Drug: Administration of methylprednisolone sodium succinate — 7-day continuous intravenous administration of methylprednisolone sodium succinate at a dose of 40mg per day
Procedure: Hyperbaric Oxygen Therapy — 1. Pressurization: It took 25 minutes to increase the pressure from 1ATA to 2.5ATA (without oxygen inhalation)
  2. Stabilization: A total of 80 minutes (30 minutes of oxygen inhalation, 5 minutes of rest, 30 minutes of oxygen inhalation, 5 minutes of rest, 10 minutes of oxygen inhalation)
  3. Decompression: 25 minutes (the first 18 minutes continued oxygen inhalation, and then 7 minutes of oxygen inhalation was stopped)
  Arms: Heperbaric oxygen-assisted Treatment

SUMMARY:
The Department of Gastroenterology plans to conduct a randomized controlled study on the efficacy analysis of hyperbaric oxygen-assisted treatment for acute severe ulcerative colitis and refractory inflammatory bowel disease. The research design is a randomized, controlled study. The objective is to compare the clinical remission rate, clinical response rate, endoscopic remission rate, and endoscopic response rate between patients with acute severe ulcerative colitis (ASUC) and refractory inflammatory bowel disease (IBD) treated with hyperbaric oxygen therapy (HBOT) as an adjuvant and those treated with standard treatment regimens. This study aims to provide clear evidence for the use of HBOT as an adjuvant treatment for ASUC and refractory IBD.

ELIGIBILITY:
Inclusion Criteria:

* According to the diagnostic criteria for ulcerative colitis in the 2018 national consensus opinion on the diagnosis and treatment of inflammatory bowel disease, it was confirmed as ulcerative colitis;
* According to the Truelove-witts standard, it was diagnosed as acute severe ulcerative colitis: the frequency of bloody stools per day is 6 times or more, and at the same time, one of the following systemic toxic manifestations is present: heart rate of 90 bpm, body temperature greater than 37.8℃, hemoglobin less than 105g/L, and erythrocyte sedimentation rate greater than 30mm/h;
* Age ≥ 18 years old;
* Patients who can and are willing to comply with the research protocol can provide a signed and dated written informed consent form.

Exclusion Criteria:

* Patients who may require immediate surgical treatment;
* Pregnant or lactating mothers;
* Patients with a score of ≥6 years old (TMM30/40/50) and <6 points in the measurement of the Eustachian tube;
* Patients with a lung bulla larger than 2 cm at the lung apex or near the pleura in the chest plain scan;
* Patients with severe liver or kidney dysfunction, heart failure or other serious systemic diseases;
* Any situation that hinders the completion of the study or interferes with the analysis of the research results, including a history of drug or alcohol abuse, a smoker who has not quit, patients with mental illness or poor compliance, those with clear immune system (including HIV infection), blood system or tumor-related diseases;
* Patients who have withdrawn their informed consent;
* Patients who have participated in other clinical trials within 3 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response | 7 days after treatment starts
  The Mayo score (or partial Mayo score) decreased by at least 3 points or more compared to the baseline (before treatment), or decreased by at least 30% from the baseline level. The single-item bleeding score decreased by at least 1 point and the absolute score was ≤ 1.

SECONDARY OUTCOMES:
Clinical remission | 7 days after treatment starts
  Mayo score total score ≤ 2 and individual score ≤ 1
Endoscopic response | 7 days after treatment starts
  The UCEIS score decreased by ≥ 2
Endoscopic remission | 7 days after treatment starts
  The UCEIS score was 0

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital of digestive diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh AK, Jha DK, Jena A, Kumar-M P, Sebastian S, Sharma V. Hyperbaric oxygen therapy in inflammatory bowel disease: a systematic review and meta-analysis. Eur J Gastroenterol Hepatol. 2021 Dec 1;33(1S Suppl 1):e564-e573. doi: 10.1097/MEG.0000000000002164. PMID 33905214
- [Background] Glover LE, Colgan SP. Hypoxia and metabolic factors that influence inflammatory bowel disease pathogenesis. Gastroenterology. 2011 May;140(6):1748-55. doi: 10.1053/j.gastro.2011.01.056. PMID 21530741
- [Background] Yamashita M, Yamashita M. Hyperbaric oxygen treatment attenuates cytokine induction after massive hemorrhage. Am J Physiol Endocrinol Metab. 2000 May;278(5):E811-6. doi: 10.1152/ajpendo.2000.278.5.E811. PMID 10780936
- [Background] Wang Y, Chen D, Chen G. Hyperbaric oxygen therapy applied research in traumatic brain injury: from mechanisms to clinical investigation. Med Gas Res. 2014 Dec 4;4:18. doi: 10.1186/2045-9912-4-18. eCollection 2014. PMID 25905012
- [Background] Memar MY, Yekani M, Alizadeh N, Baghi HB. Hyperbaric oxygen therapy: Antimicrobial mechanisms and clinical application for infections. Biomed Pharmacother. 2019 Jan;109:440-447. doi: 10.1016/j.biopha.2018.10.142. Epub 2018 Nov 3. PMID 30399579
- [Background] Chen L, Wang Y, Zhou H, Liang Y, Zhu F, Zhou G. The new insights of hyperbaric oxygen therapy: focus on inflammatory bowel disease. Precis Clin Med. 2024 Jan 18;7(1):pbae001. doi: 10.1093/pcmedi/pbae001. eCollection 2024 Mar. PMID 38344218
- [Background] Parigi TL, D'Amico F, Abreu MT, Dignass A, Dotan I, Magro F, Griffiths AM, Jairath V, Iacucci M, Mantzaris GJ, O'Morain C, Reinisch W, Sachar DB, Turner D, Yamamoto T, Rubin DT, Peyrin-Biroulet L, Ghosh S, Danese S. Difficult-to-treat inflammatory bowel disease: results from an international consensus meeting. Lancet Gastroenterol Hepatol. 2023 Sep;8(9):853-859. doi: 10.1016/S2468-1253(23)00154-1. Epub 2023 Jul 6. PMID 37423233
- [Background] De Cristofaro E, Salvatori S, Marafini I, Zorzi F, Alfieri N, Musumeci M, Calabrese E, Monteleone G. Long-Term Risk of Colectomy in Patients with Severe Ulcerative Colitis Responding to Intravenous Corticosteroids or Infliximab. J Clin Med. 2022 Mar 18;11(6):1679. doi: 10.3390/jcm11061679. PMID 35330005
- [Background] TRUELOVE SC, WITTS LJ. Cortisone in ulcerative colitis; final report on a therapeutic trial. Br Med J. 1955 Oct 29;2(4947):1041-8. doi: 10.1136/bmj.2.4947.1041. No abstract available. PMID 13260656
- [Background] Gupta V, Mohsen W, Chapman TP, Satsangi J. Predicting Outcome in Acute Severe Colitis-Controversies in Clinical Practice in 2021. J Crohns Colitis. 2021 Jul 5;15(7):1211-1221. doi: 10.1093/ecco-jcc/jjaa265. PMID 33388777
- [Background] Wehkamp J, Gotz M, Herrlinger K, Steurer W, Stange EF. Inflammatory Bowel Disease. Dtsch Arztebl Int. 2016 Feb 5;113(5):72-82. doi: 10.3238/arztebl.2016.0072. PMID 26900160
- [Result] Dulai PS, Buckey JC Jr, Raffals LE, Swoger JM, Claus PL, O'Toole K, Ptak JA, Gleeson MW, Widjaja CE, Chang JT, Adler JM, Patel N, Skinner LA, Haren SP, Goldby-Reffner K, Thompson KD, Siegel CA. Hyperbaric oxygen therapy is well tolerated and effective for ulcerative colitis patients hospitalized for moderate-severe flares: a phase 2A pilot multi-center, randomized, double-blind, sham-controlled trial. Am J Gastroenterol. 2018 Oct;113(10):1516-1523. doi: 10.1038/s41395-018-0005-z. Epub 2018 Feb 16. PMID 29453383